CLINICAL TRIAL: NCT00586872
Title: Endoscopic Mucosal Resection in Barrett's Esophagus
Brief Title: Endoscopic Mucosal Resection (EMR) in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Other Study IDs: 07-007063
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Barrett's Esophagus; Early Esophageal Adenocarcinoma
Keywords: Endoscopic Mucosal Resection
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with barretts esophagus and/or early esophageal adenocarcinoma who have undergone endoscopic mucosal resection

SUMMARY:
Existing records will be reviewed to evaluate the predictors of complications including stricture formation, bleeding or perforation associated with endoscopic mucosal resection

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a complication of gastroesophageal reflux disease in which the normal squamous lining of the esophagus is replaced by specialized columnar epithelium.1 Approximately 5%-10% of patients diagnosed with BE are thought to be at risk of developing esophageal adenocarcinoma.2 Patients with high-grade dysplasia (HGD) on biopsy are at the greatest cancer risk³. EMR is being performed clinically in our Barrett's Esophagus Unit on a regular basis during endoscopy for patients with Barrett's Esophagus and/or early esophageal adenocarcinoma. There are two predominant endoscopic mucosal resection (EMR) techniques exist using FDA approved devices - the EMR cap method using a transparent cap/snare combination and the endoscopic variceal ligation method using a band ligator/snare combination to resect tissue.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's Esophagus Early Esophageal Adenocarcinoma History of Endoscopic Mucosal Resection

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have had endoscopic mucosal resection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-10; Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Number and types of adverse events in participants who have undergone endoscopic mucosal resection with documented adverse events will be evaluated for predictors of complications | 3 months after EMR procedure
  analysis

CONTACTS AND LOCATIONS:
Overall Officials: Cadman Leggett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials